CLINICAL TRIAL: NCT00153881
Title: Docetaxel and Carboplatin Followed by a Dose-Ranging Study of Oral Capecitabine, Weekly Docetaxel, and Concomitant External Beam Radiotherapy for the Treatment of Patients With Stage II-III Carcinoma of the Esophagus and Gastro-Esophageal Junction
Brief Title: Docetaxel and Carboplatin Followed by Oral Capecitabine, Docetaxel and Radiation for Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Sanofi (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-9939; NCT00014417 (obsolete NCT alias)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal Cancer; Trimodality; Capecitabine; Xeloda; Gastro-esophageal Neoplasm; Carcinoma of the Esophagus
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Capecitabine; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Docetaxel/Carboplatin every 3 weeks for 2 cycles then concommitant chemotherapy and radiation Docetaxel weekly for 5 doses without premedication, then Capecitabine will be given orally, one dose prior to each fraction or irradiation (28 cycles).
  Interventions: Drug: Capecitabine (Xeloda)

INTERVENTIONS:
Drug: Capecitabine (Xeloda) — Neoadjuvant Chemotherapy:
  Docetaxel every 3 weeks for 2 cycles Carboplatin every 3 weeks for 2 cycles with prophylactic antibiotics and antiemetics as needed.
  Concomitant chemotherapy and radiation:
  Docetaxel weekly for 5 doses without premedication Capecitabine orally, one dose prior to each fraction of irradiation (28 cycles).
  Other Names: Capecitabine; Carboplatin; Docetaxel

SUMMARY:
The primary objective is to determine the maximum tolerated dose of oral capecitabine, in combination with fixed doses of weekly docetaxel, and concurrent thoracic radiation for the treatment of patients with clinical stage II-III cancer of the esophagus and gastroesophageal junction.

DETAILED DESCRIPTION:
This dose-ranging trial is designed to establish the phase II dose of capecitabine that can safely be given with docetaxel and radiation therapy for the treatment of patients with cancer of the esophagus and gastroesophageal junction. The docetaxel dose of 15 mg/m2/week, 5-fluorouracil dose of 200 mg/m2/week, and 50.4 Gy of thoracic radiation has been found to be the recommended doses from our initial phase I trial (DMS D9724). The Phase I study has been modified in an attempt to improve the pathological complete response rate by increasing the 5-fluorouracil exposure during thoracic radiation by replacing it with oral capecitabine. Capecitabine generates 5-fluorouracil selectively in tumor cells. This sequentially designed study of EUS staging, molecular analysis, neoadjuvant chemotherapy, concomitant chemotherapy and radiation, and surgical resection continues to expand our collaborative experience at Dartmouth Hitchcock in the treatment of cancer of the esophagus and gastroesophageal junction.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal or gastroesophageal junction cancer that is locally advanced and surgically resectable (stage II or III disease).
* No prior therapy.
* Adequate organ function.

Exclusion Criteria:

* Evidence of metastasis (celiac axis lymph nodes are allowed).
* Cervical esophageal tumors.
* Peripheral or auditory neuropathy grade >= 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2000-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of oral capecitabine in combination with fixed doses of weekly docetaxel and concurrent radiation for the treatment of patients with clinical stage II-III cancer of the esophagus and gastroesophageal junction. | Enrollment of first subject to accural of last subject/ and data analysis

SECONDARY OUTCOMES:
To determine clinical and pathological response rate, rate of resectability, duration of response, and patterns of failure for patients with esophageal and gastroesophageal junction cancers. | Enrollment of first subject to accrual of last subject/ data analysis
To determine the reliability of clinical staging and antitumor response rate assessment using endoscopic ultrasound. | Enrollment of first subject to accrual of last subject/ data analysis of study.
To investigate the feasibility of assaying thymidine phosphorylase, cyclin B, MPM-2, and perturbations in cell cycle as potential markers of efficacy. | Enrollment of first subject to accrual of last/ data analysis of study.

CONTACTS AND LOCATIONS:
Overall Officials: James R Rigas, MD, Principal Investigator — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States